CLINICAL TRIAL: NCT00027664
Title: Interferon Alpha In Combination With Thalidomide In The Treatment Of Metastatic Renal Cell Carcinoma A Randomized Phase II Study
Brief Title: Interferon Alfa With or Without Thalidomide in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ICRF-C00.204; CDR0000069055 (Registry Identifier: PDQ (Physician Data Query)); EU-20129
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-03

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; Thalidomide

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: thalidomide

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. It is not yet known if interferon alfa is more effective with or without thalidomide in treating metastatic kidney cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of interferon alfa with or without thalidomide in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of interferon alfa and thalidomide in patients with metastatic renal cell carcinoma.
* Compare the relative toxicity of interferon alfa with or without thalidomide in these patients.
* Assess the antiangiogenic effect of thalidomide by monitoring the angiogenesis-associated factors in these patients.
* Compare, in a preliminary manner, the efficacy of interferon alfa with or without thalidomide in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive interferon alfa subcutaneously 3 times a week and oral thalidomide once daily for 12 weeks.
* Arm II: Patients receive interferon alfa only as in arm I. Treatment in both arms repeats every 12 weeks in the absence of disease progression or unacceptable toxicity. Patients in arm II who develop disease progression discontinue interferon alfa and receive thalidomide only as in arm I.

Quality of life is assessed at baseline and then every 3 weeks during each study course.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma
* Measurable progressive disease, defined as non-irradiated marker lesions greater than 1 cm

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT less than 5 times ULN

Renal:

* Creatinine clearance greater than 50 mL/min OR
* Edetic acid clearance greater than 40 mL/min

Cardiovascular:

* No unstable angina or myocardial infarction within the past 6 months

Other:

* No other prior invasive malignancy except cervical intraepithelial neoplasia or nonmelanomatous skin cancer
* No chronic neurological disease causing peripheral neuropathy
* No diabetes mellitus
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least one highly effective method and at least one additional effective method of contraception for female patients and barrier contraception for male patients for at least 2 weeks before and during study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon alfa for metastatic renal cell carcinoma

Chemotherapy:

* No prior systemic chemotherapy for metastatic renal cell carcinoma
* No concurrent cytotoxic therapy

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* Concurrent local radiotherapy for symptomatic secondary sites of disease allowed if these sites are not being used as markers of disease response

Surgery:

* Not specified

Other:

* No other prior systemic treatment for metastatic renal cell carcinoma
* No concurrent chronic medication known to cause peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2001-02

PRIMARY OUTCOMES:
Safety
Toxicity
Response rate
Anti-angiogenic effect
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adrian L. Harris, MD, Study Chair — Oxford University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland